CLINICAL TRIAL: NCT01100762
Title: Can Transcranial Direct Current Stimulation (tDCS)Modulate Protective Stepping and Gait Performance of People With Parkinson's Disease
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Gad Alon, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040670
Record Dates: First submitted 2010-03-19; First posted 2010-04-09 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Cranial Electric Stimulation; Gait
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group (Experimental): 10 subjects with Parkinson's Disease receiving tPCS during the first session, treadmill walk, 7-10 days later (second session, and combined tPCS and treadmill 7-10 days week later (third session)
  Interventions: Device: Cranial Electric Stimulation (CES); Device: Treadmill; Device: CES and Treadmill

INTERVENTIONS:
Device: Cranial Electric Stimulation (CES) — We will follow the procedure described by several investigators as safe and effective. The participant will sit on a standard chair. Two commercially available surface electrodes will be embedded in an elastic head cup. Each electrode will be covered with a water soaked absorbent fabric. One positive (+) electrode will be placed over the primary motor cortex (M1) and pre-motor areas. One negative (-) electrode will be placed over the skin overlying the contra lateral supra-orbital region. The electrodes will be connected via 2 leads to a battery powered direct current stimulator. The stimulator will be programmed to deliver 0.975mA (peak 4mA) over 20 minutes.
Device: Treadmill — The participant will walk on a treadmill for 20 minutes at the individually self-selected velocity determined at baseline.
Device: CES and Treadmill — Participants will have a combined session with CES while walking on the treadmill for 20 minutes at the individually self-selected velocity determined at baseline.

SUMMARY:
The use of low level electrical stimulation when applied over the head, also called transcranial direct current stimulation (tDCS), is being tested by several groups of researchers to see if tDCS can improve movements of persons with damage to the brain. The safety and potential benefits of tDCS to children or adults patients who are paralyzed because of brain damage are reported in the medical literature. In addition, some patients with Parkinson's disease (PD) experience improvement in memory and report better use of the hand after tDCS. The treatment requires putting electrodes (pads) over the head and sending very small amount of electrical current that the patient may feel as "little tingling". Application of tDCS takes 20 min. In this study we wish to test if tDCS application can improve stepping and walking ability of subjects with PD and if the improvement is the same as when walking on treadmill. We plan to test the subject's ability to step when pulled by a laboratory testing system and also test his/her walking ability. There will be 3 sessions 7 days apart. In the first session the subject will be tested then treated for 20 min with tDCS and then tested again. In the second session the subject will be tested then walk on a treadmill for 20 min then tested again. In the third session the subject will be tested then walk on the treadmill for 20 min while receiving also tDCS and tested one last time at the end of the session. Each session will take between 2 and 3 hours.

DETAILED DESCRIPTION:
Recent advances in non-invasive electrical stimulation technology including transcranial direct current stimulation (tDCS) have provided novel and low risk options to rehabilitate the impaired ability of the central nervous system (CNS) to process sensorimotor information. Furthermore, tDCS appears to enhance CNS connectivity and there is preliminary evidence indicating that patients with Parkinson's Disease (PD) may experience improvement in working memory, the Unified Parkinson's Disease Rating Scale, simple reaction time and the Purdue Pegboard test. tDCS is inexpensive, portable and available for repeated home use. It may provide long-lasting enhancement of cortical activity in part because tDCS is easy to administer frequently and to combine it with other rehabilitation approaches including posture and gait training. However to date, no study has examined quantitatively the effects of tDCS on posture control and walking ability in patients with PD. As a first step we plan to identify the immediate effects of tDCS, as well as the added value of tDCS to treadmill exercise training, to improve posture and gait of individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult onset of PD
* A history of freezing of gait (FOG) as evidence by clinical assessment
* A stable regimen of anti-parkinsonian medications
* Ability to walk at least 10m without assistance
* Ability to walk on a treadmill for 20 minutes
* Personal weight of less than 500 Lb (because the suspension harness over the treadmill is limited to 500 Lb
* Stage 3 of the Hoehn and Yahr disability scale
* A score of >24 on the Mini Mental State Examination

Exclusion Criteria:

* Evidence of any clinically significant functional impairment related to cardiovascular, pulmonary, metabolic, other neurologic or musculoskeletal disease criterial that would preclude participation in training
* Any medical condition that might require other medical or surgical treatment during the study period
* A history of brain surgery or placement of a deep brain stimulator
* Dyskinesias > grade 2 on the Unified Parkinson's Disease Rating Scale (UPDRS)
* Any uncorrected vision or hearing problems that may limit daily activities or communication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gad Alon, PhD, PT, Principal Investigator — University of Maryland, Baltimore; Mark W Rogers, PhD, PT, Principal Investigator — University of Maryland, Baltimore; Lisa Shulman, MD, Principal Investigator — Univeristy of Maryland, Baltimore
Locations (1):
- PTRS Research Lab, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited via phone call or in person from the University of Maryland, Baltimore's Department of Neurology and the Department of Physical Therapy & Rehabilitation Sciences databases. The recruitment period was from January 2010 through June 2011.
Groups:
- Single Group: In week one, the intervention consisted of a 20 minute session of Cranial Electric Stimulation (CES). The CES dosage: the CES delivered 0.965 mA at a frequency of 5,625 pulses per second given for 20 minutes.
  In week two, the intervention was a 20 minute session walking on a treadmill. The treadmill dosage: walking at the individual subject's preferred speed on the treadmill for 20 minutes.
  In week three, the intervention was the application of CES while walking on the treadmill for 20 minutes. The CES and treadmill dosage: subjects used a combination of CES and treadmill using the same dosage of the previous two intervention sessions.
Period: Overall Study
Arm/Group | Single Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Stride Length
Description: Stride Length was measured in centimeters
Time Frame: Data collection occurred before and immediately after each training session
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Cranial Electric Stimulation (CES): In week one, the intervention consisted of a 20 minute session of Cranial Electric Stimulation (CES). The CES dosage: the CES delivered 0.965 mA at a frequency of 5,625 pulses per second given for 20 minutes.
- Treadmill: In week two, the intervention was a 20 minute session walking on a treadmill. The treadmill dosage: walking at the individual subject's preferred speed on the treadmill for 20 minutes.
- CES and Treadmill: In week three, the intervention was the application of CES while walking on the treadmill for 20 minutes. The CES and treadmill dosage: subjects used a combination of CES and treadmill using the same dosage of the previous two intervention sessions.
Arm/Group | Cranial Electric Stimulation (CES) | Treadmill | CES and Treadmill
Number analyzed (Participants) | 10 | 10 | 10
cm
  Pre Intervention | 102.10 (24.40) | 112.30 (27.30) | 109.80 (25.40)
  Post Intervention | 111.20 (22.10) | 110.40 (26.40) | 110.20 (26.70)

2. Primary Outcome: Gait Velocity
Description: Gait Velocity was measured in meters per second
Time Frame: Data collection occurred before and immediately after each training session
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Cranial Electric Stimulation (CES) | Treadmill | CES and Treadmill
Number analyzed (Participants) | 10 | 10 | 10
m/s
  Pre Intervention | 0.90 (0.23) | 102.10 (27.70) | 100.00 (24.10)
  Post Intervention | 0.985 (0.19) | 97.90 (25.80) | 98.30 (27.00)

3. Primary Outcome: Cadence
Description: Cadence was measured in steps per minute
Time Frame: Data collection occurred before and immediately after each training session
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Cranial Electric Stimulation (CES) | Treadmill | CES and Treadmill
Number analyzed (Participants) | 10 | 10 | 10
steps/min
  Pre Intervention | 106.20 (11.60) | 109.30 (10.80) | 110.00 (11.40)
  Post Intervention | 107.00 (9.80) | 107.00 (12.70) | 107.20 (10.40)

4. Primary Outcome: Number of Steps to Regain Balance
Description: Steps to regain balance were measured by the number of steps needed to recover standing balance. The steps were counted using a custom software of the motion capture system.
Time Frame: Data collection occurred before and immediately after each training session
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Cranial Electric Stimulation (CES) | Treadmill | CES and Treadmill
Number analyzed (Participants) | 10 | 10 | 10
steps
  Pre Intervention | 2.22 (1.15) | 2.00 (0.90) | 2.28 (1.31)
  Post Intervention | 2.02 (1.02) | 2.10 (1.01) | 1.94 (1.05)

5. Primary Outcome: First Step Length
Description: First step length was measured in meters from the starting position of the foot to the maximum displacement of the foot after the first step. Measurements were taken separately for forward and backward first step.
Time Frame: Data collection occurred before and immediately after each training session
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Cranial Electric Stimulation (CES) | Treadmill | CES and Treadmill
Number analyzed (Participants) | 10 | 10 | 10
m
  Pre Intervention | 0.340 (0.119) | 0.333 (0.144) | 0.316 (0.136)
  Post Intervention | 0.317 (0.126) | 0.353 (0.151) | 0.326 (0.125)

6. Primary Outcome: First Step Velocity
Description: First step velocity was measured in meters per second
Time Frame: Data collection occurred before and immediately after each training session
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Cranial Electric Stimulation (CES) | Treadmill | CES and Treadmill
Number analyzed (Participants) | 10 | 10 | 10
m/sec
  Pre Intervention | 0.859 (0.274) | 0.839 (0.369) | 0.767 (0.298)
  Post Intervention | 0.807 (0.342) | 0.873 (0.362) | 0.799 (0.275)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
1. The absence of a placebo CES
2. Limiting the stimulation to only one region of interest (Right M1)
3. Non-random order of intervention
4. CES for only one 20 minute session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No